CLINICAL TRIAL: NCT03580226
Title: Glycated Hemoglobin Targets and Glycemic Control: Link With Lipid, Uric Acid and Kidney Profile in Indonesian Diabetic Patients
Brief Title: Glycated Hemoglobin Targets and Glycemic Control in Indonesian Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Tarumanagara University (Other)
Collaborators: Hermina Podomoro Hospital (Unknown)
Responsible Party: Principal Investigator, Anthony Paulo Sunjaya, Principal Investigator, Tarumanagara University
Other Study IDs: APS001
Record Dates: First submitted 2018-06-22; First posted 2018-07-09 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Glycemic control; Lipid profile; Kidney profile; Uric acid
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Good glycemic control: Good glycemic control is defined according to the American Diabetes Association and the Indonesian Association of Endocrinologists (PERKENI) cut off of HbA1c < 7.0.
  Interventions: Other: No intervention
- Poor glycemic control: Poor glycemic control is defined according to the American Diabetes Association and the Indonesian Association of Endocrinologists (PERKENI) cut off of HbA1c >= 7.0.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study aims to compare uric acid, lipid, and kidney profile along with management and complications of Indonesian diabetic patients with good and poor glycemic control based on glycated hemoglobin profile.

DETAILED DESCRIPTION:
Adult patients (≥ 18 years of age) with type 2 diabetes which are diagnosed under ICD-10 coding of E-11 were included in this study. The inclusion criteria are patients with primary diagnosis of E11and have visited the clinic at least twice with a complete record of glucose, uric acid, lipid and kidney profile. Participants were grouped into 2 groups - good and poor glycemic control based on their glycated hemoglobin (HbA1c) levels. Good glycemic control is defined according to the American Diabetes Association and the Indonesian Association of Endocrinologists (PERKENI) cut off of HbA1c < 7.0.

Data such as age, sex, ethnic, education, BMI, glucose, uric acid, lipid, and kidney profile as well as comorbidities and type of drug used were collected from the patients' medical records. Comorbid conditions were defined as either concomitant hypertension, dyslipidemia, chronic kidney disease, hyperuricemia, or combinations of them as diagnosed in the medical records. Diabetic complications of interest include macrovascular (heart disease, stroke), microvascular (nephropathy, retinopathy, neuropathy) and a combination of both as well as infection (urinary tract infection, pneumonia). These complications were also based on the medical records. Management modalities included were lifestyle modification, use of oral antidiabetic medications or insulin, or both.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 2 Diabetes
* Must have visited the clinic at least twice, one before and one post-therapy

Exclusion Criteria:

* Type 1 Diabetes, Gestational Diabetes and other secondary diabetes types
* Unavailability of HbA1c results - pre and post-therapy
* Incomplete records of glucose, uric acid, lipid and kidney profile, comorbidities and management.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients (≥ 18 years of age) with type 2 diabetes which are diagnosed under ICD-10 diagnosis of E-11.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Lipid Profile | Through study completion, an average of 1 year
  Low-density lipoprotein (LDL), high-density lipoprotein (HDL), total cholesterol and triglyceride levels.
Kidney Profile | Through study completion, an average of 1 year
  Urea, Creatinine levels and Proteinuria
Uric Acid | Through study completion, an average of 1 year
  Uric Acid Levels

OTHER OUTCOMES:
Comorbidities | Through study completion, an average of 1 year
  Comorbid conditions were defined as either concomitant hypertension, dyslipidemia, chronic kidney disease, hyperuricemia, or combinations of them. Diabetic complications of interest include macrovascular (heart disease, stroke), microvascular (nephropathy, retinopathy, neuropathy) and a combination of both as well as infection (urinary tract infection, pneumonia).
Management | Through study completion, an average of 1 year
  Management modalities included were lifestyle modification, use of oral antidiabetic medications or insulin, or both.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Sunjaya, Principal Investigator — Tarumanagara University

IPD SHARING:
Plan to Share IPD: Undecided